CLINICAL TRIAL: NCT06610253
Title: Evaluation of the Impact of the Consumption of Plant-derived Protein Supplements Compared to Animal-derived Proteins and in Relation to the Metabolic State and Body Composition of People Practicing Physical Activity.
Brief Title: Evaluation of the Impact of the Consumption of Plant-derived Protein Supplements Compared to Animal-derived Proteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Bartosz Kroplewski, MSc Eng., University of Warmia and Mazury in Olsztyn
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 4/2023
Record Dates: First submitted 2024-05-06; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-05

CONDITIONS: Nutrition, Healthy; Body Weight Changes
Keywords: protein; physical activity; pea protein; rice protein; whey protein; plant-derived protein
MeSH Terms: conditions — Body Weight Changes; Motor Activity | interventions — Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Whey protein (Active Comparator): Healthy men engaged in physical activity. Daily supplementation with the indicated protein preparation for a period of 8 weeks. Whey group receiving 30g of a preparation containing 80% whey protein concentrate
  Interventions: Dietary Supplement: Protein
- Pea protein (Experimental): Healthy men engaged in physical activity. Daily supplementation with the indicated protein preparation for a period of 8 weeks. Pea group receiving 30g of a preparation containing 80% pea protein isolate
  Interventions: Dietary Supplement: Protein
- Rice protein (Experimental): Healthy men engaged in physical activity. Daily supplementation with the indicated protein preparation for a period of 8 weeks. Rice group receiving 30g of a preparation containing 80% rice protein isolate
  Interventions: Dietary Supplement: Protein
- MIX protein (Experimental): Healthy men engaged in physical activity. Daily supplementation with the indicated protein preparation for a period of 8 weeks. MIX group receiving 30g of a preparation containing 80% rice and pea protein isolate.
  Interventions: Dietary Supplement: Protein

INTERVENTIONS:
Dietary Supplement: Protein — Controlled, randomized, single-blind, parallel-group, prospective. Planned, parallel, randomized, single-blind, controlled clinical trial (RCT). Participants will be randomly assigned to one of four interventions: Whey Protein Concentrate - WPC, Pea Protein Isolate - PPI, Rice Protein ISOLATE - RPI, a combination of PPI and RPI to see if the intervention works together in synergy.
  The experiment was scheduled for week 8. Each participant will consume 30g of a dedicated preparation every day for 8 weeks. The planned measurements will be performed three times - before the experiment begins, after 4 and 8 weeks.

SUMMARY:
The goal of the study is to evaluate how the consumption of plant-based protein supplements compares to animal-based protein supplements in terms of their effects on metabolic state and body composition in individuals who engage in physical activity.

The increasing awareness of the health advantages of plant-based foods and the rising number of health-conscious consumers are driving the demand for plant-based supplements. Furthermore, there is a tendency for consumers to favor vegetable proteins over animal proteins.

The effect of total protein intake and its various sources on gains in lean body mass and strength in response to resistance training has been extensively studied. However, most research has focused on comparing soy protein preparations to animal-derived preparations, primarily whey protein and casein. Studies suggest that whey protein, which has a higher leucine content, may stimulate muscle protein synthesis more effectively than soy and casein. It is unclear to what extent the type of protein supplement affects strength and lean body mass in studies lasting six weeks or longer. Pea and rice proteins may be suitable replacements for highly allergenic soy protein. Consequently, there is a need for research to assess the impact of these products on human metabolic state and overall health and well-being.

DETAILED DESCRIPTION:
Dietary supplements are commonly used foodstuffs. For a long time, supplements were used mainly by people practicing sports professionally. An increasing number of supplements are dedicated to people for whom sport comes down to health-promoting physical activity. At the same time, cultural, ethical, and environmental trends encourage society to reduce animal products and use plant-based alternatives. The size of the global dietary supplement market was valued at USD 151.9 billion in 2021. It is projected to grow at an average annual rate (CAGR) of 8.9% between 2022 and 2030. Forecasts assume that consumer demand for protein supplements and amino acid products, such as creatine, tyrosine, and citrulline, will guarantee the segment of proteins and amino acids the highest share in CAGR at the level of 13.4%.

Such a dynamic trend brings with it several questions that pose new challenges to the world of science. Can protein products of plant origin compete with the preparations based on proteins of animal origin, which have been present for many years? What effects can the investigators expect from systematic supplementation of vegetable proteins? Which of the vegetable proteins is the best substitute for proteins of animal origin, and does supplementation with vegetable proteins carry no additional risks? In the study, the investigators want to compare four protein preparations: whey protein, pea protein, rice protein, and a preparation composed of pea and rice protein mixed in the right proportion to increase its biological value by complementing the limiting amounts of amino acids. Pea and rice proteins may be a promising replacement for highly allergenic proteins such as soy protein. Therefore, there is a need to research the assessment of the impact of these products on the metabolic state of humans in terms of health and quality of life.

Another research aspect regarding the consumption of proteins of various origins is the assessment of their impact on the intestinal microbiota profile. In recent years, the number of scientific publications on the role of intestinal microbiota in shaping human health has been increasing. It is now known that the intestinal microbiota is not only involved in the processes related to the digestion and absorption of nutrients. Bacteria included in the intestinal microbiota perform various functions, and their proper quantitative and qualitative structure supports the homeostasis of the whole organism, shaping immunity, metabolism, and the synthesis of many chemical compounds.

Research hypotheses:

1. Protein preparations of vegetable origin (rice protein isolate, pea protein isolate) when covering the demand for leucine (protein from food + preparation) will not show significant differences in body composition compared to a protein preparation of animal origin (WPC).
2. The combination of the intervention with the preparations (pea and rice proteins), due to the reduction in the amount of limiting amino acids, will have a more favorable effect on the total protein utilization than the separate intervention with the preparation of rice protein and pea protein.
3. Increased protein supply will help reduce muscle mass loss during intense physical exercise.
4. A diet enriched with a protein preparation affects the biochemical parameters of the blood and the microbiota profile.

2. Importance of the project Resistance exercise is widely regarded as a key strategy in developing muscle mass, strength, and endurance. They are also an effective tool in limiting the progression of sarcopenia. Research shows that resistance training alone may not be enough. Stimulation of protein synthesis by resistance exercise also depends on protein supply . Protein intake greater than the RDA is beneficial in maintaining lean mass during periods of intense exercise or controlled weight loss.

The biological value of protein goes beyond its amino acid composition and digestibility. In healthy individuals, the slow release of amino acids into the portal vein and then into the systemic circulation in response to bolus protein intake improves nitrogen retention and reduces urea production. In addition, the protein is a source of essential amino acids (EAAs), of which branched-chain amino acids (BCAAs) are associated with the stimulation of skeletal muscle protein synthesis. Studies show that whey proteins achieve better nitrogen retention than soy or casein, which is probably due to the high content of essential amino acids (especially leucine). However, leucine consumption above 3.5g per day does not seem to provide additional benefits.

The interest of the clinical and consumer market is increasingly focused on the use of protein supplements as dietary ingredients to maintain or increase skeletal muscle mass. Recent studies suggest that the consumption of plant-derived proteins (soy and wheat proteins) causes a weaker reaction of muscle protein synthesis compared to animal-derived proteins. The weaker anabolic properties of plant proteins can be attributed to lower digestibility and a greater synthesis of urea from plant-derived amino acids compared to animal-derived proteins. The latter may be related to plants' relative lack of certain essential amino acids. In addition, most plant proteins are relatively low in leucine, which may further reduce their anabolic properties. The literature data show that proteins of plant origin can support the reduction of excessive body weight and lower the level of lipids in the blood. They can also positively affect kidney and liver function. Research to date has focused mainly on plant proteins derived from soy and wheat, therefore there is a need to thoroughly investigate the effects of plant protein preparations other than soy and wheat.

Selection of protein preparations and justification

The investigators selected 4 protein preparations for the study:

1. - whey protein concentrate (WPC) with a protein content of 80%
2. - rice protein in the form of an isolate (RPI) with a protein content of 80%
3. - pea proteins in the form of an isolate (PPI) with a protein content of 80%
4. - a preparation combining RPI and PPI in a 1 to 1 ratio (MIX) with a protein content of 80, created for the study

Description of the proteins selected for the study:

Whey proteins are distinguished by fast digestion and high content of essential amino acids (EAA), which are necessary to stimulate skeletal muscle protein synthesis. In terms of amino acid composition, whey is similar to muscle proteins. Whey has the highest level of BCAAs. It is the most commonly used protein supplement among athletes and people practicing physical activity. It plays an important role in protein synthesis, increasing lean muscle mass and in the metabolism of carbohydrates that provide energy during exercise, thus improving athletic performance.

Rice proteins - until recently, rice flour was mainly processed by industry to collect starch residues, and proteins used for animal feed. Nowadays, rice proteins are considered by producers as valuable raw materials. The protein content of rice can vary depending on genotype, climate, and cultivation practice, but is typically 7-10% of the weight of the grain. Rice protein is becoming an increasingly popular alternative to animal proteins. It contains all essential amino acids and has hypoallergenic properties. Thanks to these properties, rice protein becomes a food ingredient with a wide range of applications in infant formulas, foodstuffs, and dietary supplements for athletes. The Protein Digestibility Corrected Amino Acid Index (PDCAAS) for rice bran protein is 0.90 and for soy protein is 0.95. These are very similar results and only slightly worse compared to whey 1.00. In addition, brown rice concentrate contains 36% EAA and 18% BCAA. Therefore, rice protein derived from brano r endosperm is a potential replacement for many animal products.

Pea proteins have a well-balanced amino acid profile with a high lysine content and achieve a PDCAAS of 0.89. Relatively low calorific value and the fact that pea proteins do not contain gluten and are a vegan product make them gain more and more recipients. They are fairly well tolerated by most people and easily digestible compared to some other sources of plant protein such as soy or beans. Pea proteins are widely used as an ingredient in food products such as protein drinks, protein powders, protein bars, cookies, and other processed foods. They can also be used as an ingredient in baked goods, soups, sauces, and salads. Studies show that pea proteins can support the process of muscle mass gain in people performing resistance training. Thanks to its availability, low cost, nutritional value, and health benefits, pea protein can be used as a new and effective alternative to soy or animal proteins in functional foods.

Various strategies can be used to improve the anabolic properties of plant proteins, these may include: enrichment of plant protein sources with amino acids, i.e. methionine, lysine, and/or leucine, consumption of more plant protein sources, consumption of multiple sources of protein in to provide a more balanced amino acid profile. Milk and vegetable protein blends achieve more balanced amino acid profiles with higher scores compared to single-component proteins. However, the effectiveness of such nutritional strategies in postprandial muscle protein synthesis requires further research.

Growing awareness of the health benefits of plant-based foods and the growing number of health-conscious consumers are key drivers of demand for plant-based supplements. Consumers are increasingly switching from animal proteins to vegetable proteins. This will likely shift consumers' predisposition towards plant-derived supplements.

Much attention has been devoted to determining the effect of total protein intake and its various sources on gains in lean body mass and strength in response to resistance training. Most studies have focused on the comparison of soy protein preparations with animal-derived preparations based mainly on whey protein and casein. Studies indicate that whey protein, probably related to the higher content of leucine, better stimulates muscle protein synthesis. This process occurs to a greater extent than in the case of proteins such as soy and casein. In 2013, a study was conducted that compared the effects of rice and whey protein on body weight composition. A study conducted for 8 weeks on 24 young men systematically performing strength training showed that there were no differences between rice protein and whey protein when covering the demand for leucine. In 2019, research results were published describing the effect of whey and pea protein supplementation on physiological adaptations after an 8-week intensive functional training. They did not show a significant difference for such parameters as body weight or body fat content after the 8-week intervention. Pea and rice proteins may be a promising replacement for highly allergenic proteins such as soy protein.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 18-40, practicing systematic physical activity at least twice a week.

Exclusion Criteria:

* food allergies to milk, pea and rice proteins.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
analysis of selected blood biochemical parameters - electrolytes (Na, K, Cl) | 3 times. at the beginning, after 4 weeks and after 8 weeks
  The measurement electrolytes (Na, K, Cl) will be performed by the MFA Analytical Laboratory in Olsztyn. Result values will be expressed in units - mmol/l
analysis of selected blood biochemical parameters - lipid profile | 3 times. at the beginning, after 4 weeks and after 8 weeks
  The measurement of lipid profile (HDL,LDL, non HDL, triglycerides) will be performed by the MFA Analytical Laboratory in Olsztyn. Result values will be expressed in units - mg/dl
analysis of selected blood biochemical parameters - liver condition | 3 times. at the beginning, after 4 weeks and after 8 weeks
  The measurement of liver condition (ASPAT, ALAT, GGTP, LDH) will be performed by the MFA Analytical Laboratory in Olsztyn. Result values will be expressed in units - U/L
analysis of selected blood biochemical parameters - protein metabolism | 3 times. at the beginning, after 4 weeks and after 8 weeks
  The measurement of serum total protein, total bilirubin, serum urea, serum creatinine, serum uric acid will be performed by the MFA Analytical Laboratory in Olsztyn. Result values will be expressed in units - mg/dl
analysis of the amino acid profile in plasma and urine samples | 3 times. at the beginning, after 4 weeks and after 8 weeks
  Analysis of the amino acid profile in plasma and urine samples of volunteers collected during the experiment will be carried out using the HPLC-MS method
analysis of the stool samples | 3 times. at the beginning, after 4 weeks and after 8 weeks
  It will be assessed by next-generation sequencing (NGS) of the bacterial specific 16S rRNA variable region. DNA will be extracted from the samples using the QIAamp Fast DNA Stool Mini Kit (Qiagen) according to the manufacturer's instructions. The extracted DNA will be used to assess the microbiota profile by amplifying the V3-V4 region of the 16S rRNA gene using primers and protocols according to the instructions for preparing the 16S metagenomic sequencing library
body composition analysis - body weight | 3 times. at the beginning, after 4 weeks and after 8 weeks
  Measurement of body composition parameters - body weight will be performed using the body scale that is part of the Body Composition Analyzer SECA (515mBCA). Body weight will be expressed in units - kilograms, with an accuracy of 0.01 kg
body composition analysis - body high | 3 times. at the beginning, after 4 weeks and after 8 weeks
  The measurement of body composition parameters - height, will be performed using a validated measure included in the Body Composition Analyzer SECA equipment (515mBCA). Participants' height will be expressed in units - meters with an accuracy of 0.01 m
body composition analysis | 3 times. at the beginning, after 4 weeks and after 8 weeks
  Measurement of body composition parameters (body fat, total body water, skeletal muscle mass, bone mass will be performed using the bioimpedance method using the Body Composition Analyzer SECA (515mBCA). Parameters will be expressed in units - kilograms, with an accuracy of 0.01 kg and their conversion into percentages of total body weight
body composition analysis - BMI | 3 times. at the beginning, after 4 weeks and after 8 weeks
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms (kg) and height in metres (m).

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Kroplewski, MSc, Eng., Principal Investigator — UWM Olsztyn; Katarzyna Przybyłowicz, Prof Eng., Study Director — UWM Olsztyn; Tomasz Sawicki, PhD, Eng., Study Director — UWM Olsztyn
Locations (1):
- University of Warmia and Mazury, Olsztyn, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No